CLINICAL TRIAL: NCT00052624
Title: A Phase I Multicenter Trial Of Intratumoral/Interstitial Therapy With HN66000, NC66000 (TransMID) In Patients Between 5 and 18 Years Of Age With Progressive Or Recurrent Glioblastoma Multiforme Or Anaplastic Astrocytoma
Brief Title: Immunotoxin Therapy in Treating Children With Progressive or Recurrent Glioblastoma Multiforme or Anaplastic Astrocytoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xenova Biomedix (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: MUSC-10550; KSB-311P/CI/001; CDR0000258574 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2004-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent childhood cerebral astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma | interventions — Tf-CRM107

INTERVENTIONS:
Biological: transferrin-CRM107

SUMMARY:
RATIONALE: Immunotoxins can locate tumor cells and kill them without harming normal cells. Immunotoxin therapy may be an effective treatment for glioblastoma multiforme and anaplastic astrocytoma.

PURPOSE: Phase I trial to study the effectiveness of immunotoxin therapy in treating children who have progressive or recurrent glioblastoma multiforme or anaplastic astrocytoma

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of intratumoral transferrin-CRM107 in pediatric patients with progressive or recurrent glioblastoma multiforme or anaplastic astrocytoma.
* Determine the safety of this drug in these patients.
* Determine the efficacy of this drug in these patients.
* Compare the efficacy of this drug in patients with different histological types of tumor, degrees of transferrin receptor expression, and serum antidiphtheria antibody titer levels.

OUTLINE: This is a dose-escalation, open-label, multicenter study. Patients are assigned to 1 of 2 treatment groups by age (5-9 vs 10-18).

All patients undergo stereotactic radiosurgery for tumor biopsy and placement of 2 intratumoral silastic infusion catheters pre-loaded with transferrin-CRM107 (Tf-CRM107).

* Group 1 (ages 5-9): Patients receive intratumoral Tf-CRM107 over 3-7 days via catheter. Treatment repeats after 6-10 weeks in the absence of unacceptable toxicity. Three cohorts of 3-6 patients receive escalating doses of Tf-CRM107 until the maximum tolerated dose (MTD) is determined.
* Group 2 (ages 10-18): Patients receive intratumoral Tf-CRM107 as in group 1. Two cohorts of 3-6 patients receive escalating doses of Tf-CRM107 until the MTD is determined.

The MTD in both groups is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed monthly for 6 months and then every 3 months for 6 months.

PROJECTED ACCRUAL: A total of 3-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme or anaplastic astrocytoma with the following tumor characteristics:

  * Unifocal
  * Unilateral and supratentorial
  * Diameter no greater than 3.5 cm by contrast-enhanced MRI
* No more than 1 satellite tumor
* Recurrent or progressive disease

  * Progressive disease defined as at least 25% increase in tumor volume by serial MRI or CT scans and/or at least 15% increase in the largest cross-sectional area of tumor as defined by the area of contrast agent enhancement
* Must have received prior conventional treatment comprising both of the following:

  * Surgery (biopsy or debulking)
  * Radiation therapy
* No evidence of mass effect on CT scan or MRI with more than a 5 mm midline shift and/or nausea, vomiting, reduced level of consciousness, or clinically significant papilledema

PATIENT CHARACTERISTICS:

Age

* 5 to 18

Performance status

* Karnofsky 60-100% OR
* Lansky Play 50-100%

Life expectancy

* At least 3 months

Hematopoietic

* Platelet count at least 100,000/mm^3
* Absolute neutrophil count at least 1,000/mm^3

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* AST and ALT no greater than 2.5 times the upper limit of normal (ULN)
* PT or aPTT no greater than 1.5 times ULN

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 2 months after study
* No acute viral, bacterial, or fungal infection requiring therapy

  * Topical treatment for oral candidiasis allowed
* No other concurrent medical condition that would preclude anesthesia

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior transferrin-CRM107

Chemotherapy

* More than 1 month since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* More than 3 months since prior biodegradable polymer wafers
* No concurrent chemotherapy

Endocrine therapy

* Must be on stable dose of steroids for 7 days prior to infusion

Radiotherapy

* See Disease Characteristics
* More than 3 months since prior radiotherapy
* More than 3 months since prior stereotactic radiosurgery
* More than 6 weeks since prior craniospinal irradiation
* No prior brachytherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* More than 1 month since prior surgery including tumor surgery or debulking
* No other concurrent surgery

Other

* More than 30 days since prior investigational agents
* No other concurrent investigational therapy
* No other concurrent anti-cancer drugs

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2002-07

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Rossi, MD, Study Chair — Xenova Biomedix
Locations (2):
- United States (2):
  - Children's Hospital of Orange County, Orange, California
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina